CLINICAL TRIAL: NCT03840694
Title: Nicotine Withdrawal and Reward Processing: Connecting Neurobiology to Real-world Behavior
Acronym: NicWith
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI leaving for another institution.
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: Pro00101055
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Cigarette Smoking; Nicotine Withdrawal
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Intervention Model Description: Participants will abstain from smoking for 24 hours before one MRI scan and continue smoking as usual before the other.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smoking Abstinence (Other): Participants will abstain from smoking for 24 hours before one MRI scan. Smoking abstinence will be confirmed using exhaled carbon monoxide breath testing
  Interventions: Other: Smoking Abstinence
- Ad Lib Smoking (Other): Participants will continue smoking as usual (i.e. "ad lib") before one MRI scan and smoke one additional cigarette immediately prior to scanning. Continued smoking will be confirmed using exhaled carbon monoxide breath testing.
  Interventions: Other: Ad Lib Smoking

INTERVENTIONS:
Other: Smoking Abstinence — Participants will abstain from smoking for 24 hours.
  Arms: Smoking Abstinence
Other: Ad Lib Smoking — Participants will continue smoking as usual (i.e. ad lib) and smoke one cigarette of their own brand immediately prior to scanning.
  Arms: Ad Lib Smoking

SUMMARY:
This study is designed to find out how smoking affects the way the brain responds to pleasure and how this impacts smokers' behavior. Participants will complete three sessions. The first session will be a screening and training visit to determine final eligibility. Eligible participants will work with a researcher to develop brief scripts about times when they smoke and do other activities. Next, participants will attend two magnetic resonance imaging (MRI) scans - one after abstaining from smoking for 24 hours and the other after smoking as usual. After the second MRI, participants will answer questions on their phone every day for two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy
* Right-handed
* Smoke >= 10 cigarettes per day
* Smoking regularly for >= 1 year
* Carbon Monoxide (CO) > 8 at screening (or urinary cotinine > 100)
* Own a compatible smartphone
* Able to read and understand English
* Able to identify at least 4 pleasurable activities they do not do concurrently with smoking or associate with smoking

Exclusion Criteria:

* Regular use of "roll your own" cigarettes
* Planning to quit smoking within the next 60 days
* Current or planned smoking cessation treatment
* Regular use of smokeless tobacco or other nicotine products
* Expired CO > 80 parts per million
* Breath alcohol > .000 at screening (re-attempts are allowed)
* Positive toxicology screen for exclusionary drugs
* Use of exclusionary medications
* Significant medical problems
* Currently breastfeeding, pregnant, or planning to become pregnant
* Enrollment in another study utilizing Spectrum cigarettes within the last 3 months
* Irregular slee-wake cycles (e.g. swing-shift work, unusual sleep patterns)

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2021-05-13 (Actual); Study Completion 2021-05-13 (Actual)

PRIMARY OUTCOMES:
Blood Oxygen Level Dependent (BOLD) Activation | Approximately 1-3 weeks
  BOLD activation in brain reward network regions
Ecological Momentary Assessment (EMA) Pleasure Ratings | 2-6 weeks
  Anticipated and actual pleasure ratings acquired each day during EMA portion of study. Individual items are based on the 12-item Tripartite Pleasure Inventory (TPI). Participants rate their anticipated pleasure for activities they expect to engage in each day using a 0 (No pleasure) to 4 (Extreme pleasure) scale in the morning. They will then rate their actual experienced pleasure for activities they actually did engage in the evening using the same scale. Scores are summed across items for a theoretical range of 0-48.

CONTACTS AND LOCATIONS:
Overall Officials: Jason A Oliver, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University School of Medicine, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Detailed protocols, datasets and additional information will be available from the Principal Investigator and research team upon request. In order to maintain compliance with the Health Insurance Portability and Accountability Act (HIPAA) requirements, as well as university data security policies, all data will be anonymized according to HIPAA guidelines prior to being shared. Individual participant scripts will not be made publicly available due to privacy concerns and because this could impact the nature of information participants were willing to provide for scripts. Data will be provided in widely accessible formats for both self-report and imaging data. We will work with the Office of Research Contracts to obtain guidance regarding any required Data Use Agreements as needed.
Supporting Information: Study Protocol
Time Frame: We anticipate making data available within 6 months of study completion. It will be available for an indefinite period of time.
Access Criteria: Contact PI for details.